CLINICAL TRIAL: NCT00174148
Title: Sensorimotor Dysfunction of Individuals With Neck Pain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701250
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2005-12-21 (Estimated); Status verified 2004-12

CONDITIONS: Posterior Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
Systematically assessing the proprioception-coordination capacity of the spine in patients with different severity of neck disability could reveal how the dysfunction of the sensory-motor system was progressed. From the result of the research, a prospective study would be designed to test the hypotheses that described the mechanism of neck pain based on the results to the present study.

DETAILED DESCRIPTION:
The purposes of this research were to investigate the effect of age and chronic neck pain on cervical proprioception, the change of ultrasonographic (USD) patterns in deep neck muscle and superficial neck muscles. The hypotheses of this research included: 1) the alteration of neck proprioception is determined predominantly by the changed activation deep neck muscles and superficial neck muscles. 2) Age factor contributes to the alteration of cervicocephalic sensibility, USD pattern of deep and superficial muscles. 3) Chronic pain contributes to the alteration of cervicocephalic sensibility, USD pattern of deep and superficial muscles.

Neck proprioception is measured by an ultrasound-based coordinate measuring system (CMS 70P, Zebris, Germany) by asking the subjects to performed head repositioning to the neutral head position or to a target position in three cardinal plane. These repositioning error expressed in root mean square errors could represent the craniocervical kinesthetic sensibility. The change of muscle thickness (mm) of the superficial (Trapezium, Splenius) and deep (semispinalis cervicis and multifidus) dorsal neck muscle is measured by a real-time ultrasonographic scanner (HDI 5000, ATL Ultrasound, USA). Image is obtained for each cervical level, and the thickness of the muscle is identified manually using a custom-written C++ computer graphic program. The measurements of pain intensity and pain frequency are modified from the symptoms questionnaire to indicate the intensity, location, frequency and duration of pain and disability of the subjects. The age and pain effects for each independent variables measured in patients with chronic neck pain (pain: intensity, location, frequency, and duration, NDI), will be tested with the General Linear Model (GLM; age and pain factors). The confounding factors such as gender, range of motion, body height and weight are controlled in the regression model.

ELIGIBILITY:
Inclusion Criteria:

* posterior neck pain with duration over 3 months

Exclusion Criteria:

* surgery on cervical spine
* achilosing spondylitis
* diabetes mellitus
* traumatic injury directly over head and neck area
* progressing neurological disease

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60
Dates: Start 2005-07; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Shwu-fen Wang, PT Phd, Study Chair — National Taiwan University Hospital
Locations (1):
- School and Graduate Institution of Physical Therapy, College of Medicine,Nnational Taiwan University, Taipei, Taiwan